CLINICAL TRIAL: NCT01364142
Title: A Blind Maneuver to Position an Endobronchial
Brief Title: A Blind Maneuver to Position an Endobronchial Blocker
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, professor, Seoul National University Hospital
Other Study IDs: JHBahk_bronchial blocker
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: One Lung Ventilation; Endobronchial Blocker; Thoracic Surgery; Fiberoptic Bronchoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- thoracic surgery: Patients undergoing thoracic surgery in which one lung ventilation is needed.
  Interventions: Procedure: endobronchial blocker

INTERVENTIONS:
Procedure: endobronchial blocker — After intubation of endotracheal tube, the Uniblocker® was inserted into the endotracheal tube and advanced step by step with inflation of the blocker balloon until the peak inspiratory pressure dropped abruptly.

SUMMARY:
One-lung ventilation can be provided by an endobronchial blocker. The Uniblocker® (Fuji Systems Corporation, Tokyo, Japan) was relatively recently introduced into clinical practice. We will try to devise a blind method to locate the Uniblocker® without the aid of fiberoptic bronchoscopy.

DETAILED DESCRIPTION:
The use of a fiberoptic bronchoscopy (FOB) appears to be fundamental to adjusting position of the bronchial blocker in the targeted mainstem bronchus. However, there can be occasions when a FOB is unavailable or inapplicable. Therefore, we will try to devise a blind method to locate the blocker without the aid of FOB in patients undergoing thoracic surgery.

After intubation of endotracheal tube (ETT), the Uniblocker® is inserted into the ETT and is advanced until the blocker balloon comes out of the ETT tip. At this time, the blocker balloon is inflated with air and the peak inspiratory pressure (PIP) will abruptly increase. And then, the blocker is rotated to the thoracotomy side and advanced to the carina step by step at 0.5 cm intervals. When the PIP drops abruptly, the blocker cuff is deflated completely and advanced to 3 cm further. The blocker cuff is inflated again. Using a FOB, the position of the blocker is recorded and we will evaluate the success rate of proper blocker position.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracic surgery who need one lung ventilation

Exclusion Criteria:

* patients who have a lesion in trachea or mainstem bronchi
* severe tracheal deviation
* patients who do not agree to informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thoracic surgery
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyon Bahk, PhD, MD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Hong DM, Seo JH, Chang Kim H, Nam K, Bahk JH. A novel maneuver to blindly position bronchial blockers. Minerva Anestesiol. 2013 Oct;79(10):1126-31. Epub 2013 May 29. PMID 23719651